CLINICAL TRIAL: NCT02037464
Title: CAPSAICIN Trial: A Prospective Study of Capsaicin in Subjects With Clinically Localized Prostate Cancer Undergoing Active Surveillance or Radical Prostatectomy
Brief Title: CAPSAICIN Trial: Assessing Capsaicin as a Chemopreventive Agent for Prostate Cancer
Acronym: CAPSAICIN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Laurence Klotz, Dr. Laurence Klotz, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 264-2013
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Active Surveillance; Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Capsaicin Supplement (Experimental)
  Interventions: Dietary Supplement: Capsaicin Supplement (Cayenne by Nature's Way)

INTERVENTIONS:
Dietary Supplement: Capsaicin Supplement (Cayenne by Nature's Way) — One capsule of the supplement to be taken twice daily.
  Other Names: Naturesway Cayenne 40,000 H.U. (NPN #80013036)

SUMMARY:
The purpose of this study is to determine the chemopreventive properties of capsaicin, the active compound in chili peppers, in prostate cancer patients enrolled in the active surveillance program or patients scheduled to undergo radical prostatectomy.

DETAILED DESCRIPTION:
Rationale A large body of evidence supports the role of dietary factors in prostate cancer development and progression. Most of this evidence suggests that diet high in fat including red meat and low in micronutrients and other anti-oxidants, increases the risk of disease. We are interested in the therapeutic potential of the dietary agent, capsaicin (CAP). Capsaicin is the active compound in chili peppers, and related plants. Pre-clinical studies have found that capsaicin has potent growth inhibitory and pro-apoptotic effects. It is thought that consumption of a capsaicin supplement may have a clinical benefit for subjects with localized prostate cancer who have chosen to be managed by active surveillance or improve surgical outcome of patients undergoing radical prostatectomy.

Objective(s) Primary • To assess the effect of capsaicin daily therapy on the expression of ki67 and p27 biomarkers in a post-treatment biopsy or prostate specimen from RP.

Secondary

* To assess the effect of therapy with repeat oral dosing of capsaicin two times daily on Prostate Specific Antigen (PSA) kinetics in men on active surveillance for localized prostate cancer
* To assess the effect of therapy with repeat oral dosing of capsaicin two times daily on grade and the presence of prostatic intraepithelial neoplasia (PIN) in a post-treatment biopsy
* To assess the effect of therapy with repeat oral dosing of capsaicin two times daily on the expression of markers of apoptosis, cell cycle, TRP-V1 and TRP-V6
* To assess the safety and tolerability of capsaicin therapy in men on active surveillance (AS) for prostate cancer
* To assess alterations in prostate volume and time to recurrence

Endpoint(s) Primary

• Determine effect of capsaicin therapy on expression of ki67 and p27 biomarkers in a post-treatment biopsy

Secondary

* Determine effect of capsaicin daily therapy on PSA kinetics in men on active surveillance for localized prostate cancer
* To evaluate the effect of capsaicin daily therapy on grade and the presence of prostatic intraepithelial neoplasia (PIN) in post treatment biopsy
* To assess the effect of capsaicin therapy on the expression of markers of apoptosis, cell cycle, TRP-V1 and TRP-V6

Safety and Tolerability

* Adverse events (AEs)
* Clinical laboratory evaluations (PSA, electrolytes, biochemistry, hematology, cholesterol)

Pharmacodynamic

* Levels of serum capsaicin (CAP)
* Levels of serum testosterone (T)

Study Design This is a phase II, open label, single centre study to evaluate the efficacy and safety of repeat oral dosing of one CAP capsules twice times daily for 6 months prior to a prostate biopsy in men on active surveillance for localized prostate cancer, as well as 6 weeks prior to radical prostatectomy (RP).

Study Population One hundred men men monitored (sixty from active surveillance (AS) and forty patients scheduled to undergo radical prostatectomy) will be eligible for participation. Subjects must satisfy all inclusion and exclusion criteria. A sufficient number will be enrolled to achieve at least 100 completed subjects

ELIGIBILITY:
Inclusion Criteria:

1. Subject is >19 years of age
2. Subject has a histologically documented diagnosis of prostate adenocarcinoma
3. Being monitored by active surveillance (see Table 1) for favourable risk prostate cancer as defined by the following:

   1. Clinical stage T1b, T1c, T2a or T2b at the time of diagnosis
   2. Clinical (diagnostic biopsy) Gleason score < 6
   3. PSA < 10.0 ng/ml (ug/L)
4. Tumour material from most recent prostate biopsy available with sample (up to 10 unstained slides) collected for determination of ki67 and p27 biomarker expression.
5. Scheduled to have an active surveillance mandated transrectal ultrasound (TRUS) guided biopsy within 6 - 12 months of Day 1 of the study

Exclusion Criteria:

1. Previous malignancy (not including curatively treated basal or squamous cell carcinoma of the skin) within the previous 5 years. (Ta bladder cancer with negative surveillance cystoscopy within the past 2 years may be included.)
2. No previous or current treatment (medical therapy or radical intervention) for prostate cancer excluding biopsy
3. Inability to undergo TRUS biopsy
4. Concurrent administration of the following medications is not permitted during the protocol:

   * 5 α-reductase inhibitors
   * Cytotoxic chemotherapy
   * Immunotherapy
   * Hormonal therapy (megestrol, medroxyprogesterone, cyproterone, diethylstilbestrol, hyrodcortisone, etc.)
   * Non-steroidal anti-androgens (bicalutamide, nilutamide, flutamide, etc.)
   * Luteinizing hormone releasing Hormone (LHRH) analogues (leuprolide, goserelin, etc.)
   * Ketoconazole
   * PC-SPES and any other preparations thought to have endocrine effects
   * Medications which inhibit cholesterogenesis ('statin' medications, etc.)
5. Eastern Cooperative Oncology Group (ECOG) Performance Status > 2
6. Known or history of liver disease (total bilirubin, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 upper limit of normal at screening visit)
7. Subject has a minimum life expectancy of < 5 years
8. Subject is unable to give written and informed consent

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-06 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Biomarker Changes | 6-8 weeks or 9 +/-3 months
  Determine effect of capsaicin therapy on expression of ki67 and p27 biomarkers in a post-treatment biopsy.

SECONDARY OUTCOMES:
PSA Kinetics | 1 year
Tumor grade | 1 year
Biomarkers | 1 year
  To assess the effect of capsaicin therapy on the expression of markers of apoptosis, cell cycle, TRP-V1 and TRP-V6

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Klotz, MD, Principal Investigator — Sunnybrook Hospital
Locations (1):
- Sunnybrook Hospital, Toronto, Ontario, Canada